CLINICAL TRIAL: NCT03841500
Title: Prospective Evaluation of Osseous Integration and Patient Outcomes In Allograft ACL Reconstruction Comparing Tightrope Versus Biocomposite Interference Screw Fixation
Brief Title: Prospective Evaluation of Osseous Integration in ACL Reconstruction Comparing Tightrope vs Interference Screw Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kelsey-Seybold Clinic (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Anup Shah, Principal Investigator, Kelsey-Seybold Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAIRB-14-0044
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: ACL - Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aperture (biocomposite screw) fixation (Active Comparator): 16 patients in this arm underwent ACL reconstruction with the allograft fixed in the femoral tunnel with a biocomposite interference screw (BioComposite Screw, Arthrex, North Naples, FL; or MILAGRO screw, DePuy Mitek, Raynham, MA, USA).
  Intervention: ACL reconstruction with the allograft fixed in the femoral tunnel with a biocomposite interference screw.
  Interventions: Device: Biocomposite intereference screw femoral tunnel fixation
- Suspensory (endobutton) fixation (Active Comparator): 17 patients in this arm underwent ACL reconstruction with the allograft secured in the femoral tunnel with a cortical button (TightRope, Arthrex, North Naples, FL, USA).
  Intervention: ACL reconstruction with the allograft secured in the femoral tunnel with a cortical button.
  Interventions: Device: Endobutton (Tightrope) femoral tunnel fixation

INTERVENTIONS:
Device: Biocomposite intereference screw femoral tunnel fixation — ACL reconstruction using biocomposite intereference screw for femoral tunnel fixation
  Arms: Aperture (biocomposite screw) fixation
Device: Endobutton (Tightrope) femoral tunnel fixation — ACL reconstruction using endobutton (Tightrope) for femoral tunnel fixation
  Arms: Suspensory (endobutton) fixation

SUMMARY:
The purpose of our study was to compare osseous integration of the bone block in Achilles tendon allograft ACL reconstruction using a cortical button versus biocomposite interference screw fixation. The primary outcome was bone block incorporation within the femoral tunnel at six months. Our null hypothesis was that there is no difference in osseous incorporation or outcome with either type of femoral fixation in primary ACL reconstruction with Achilles tendon allograft. Our secondary outcomes were pain and clinical outcome scores between the two groups.

DETAILED DESCRIPTION:
After obtaining institutional review board approval the investigators conducted this prospective randomized controlled trial with goal of 1:1 allocation ratio between the two study groups. All subjects were recruited at the preoperative appointments. The senior investigator discussed ACL reconstruction with the patients. Appropriate preoperative counseling was performed regarding graft options. If inclusion criteria were met, patients received information about the study. Informed consent was obtained from those choosing to enroll in the study including consent for a CT scan at the six month postoperative time period. The patients were randomized for fixation technique on the day of surgery from a list using the medical record number. Patients underwent ACL reconstruction with Achilles tendon allograft with femoral-sided bone block fixation with either (1) a biocomposite interference screw (aperture fixation) or (2) cortical button (suspensory fixation).

The inclusion criteria included patients between the ages of 18 and 50 able to provide informed consent with ACL tears meeting the indications for reconstruction and electing to undergo reconstruction with an Achilles tendon allograft. Excluded patients included those with a history of prior ACL reconstruction, pregnancy, inflammatory disease, a primary bone disorder, those taking bone resorption inhibitor medications, and those with injuries to the collateral ligaments or posterior cruciate ligament.

All surgeries were performed by a single surgeon at a single institution using the same technique. Initial diagnosis of ACL deficiency was made on physical exam and magnetic resonance imaging. This was confirmed with arthroscopy at the beginning of the case. The Achilles-calcaneal bone allograft was thawed. The tendinous portion was tubularized and whip-stitched with a locking Fiberloop suture (Arthrex, North Naples, FL, USA). Sutures were passed through the bone block and the graft diameter was measured. The graft was then pre-tensioned. Femoral tunnels were made using the anteromedial portal at 120 degrees of knee flexion. The tibial tunnel was created using an outside-in technique over a pin centered at the ACL footprint. In the aperture fixation group, the bone graft end was pulled through into the femoral tunnel and secured with a biocomposite interference screw (BioComposite Screw, Arthrex, North Naples, FL; or MILAGRO screw, DePuy Mitek, Raynham, MA, USA). In the suspensory fixation group, a cortical button (TightRope, Arthrex, North Naples, FL, USA) was pulled through the femoral cortex and used to shuttle the Achilles bone plug into the femoral tunnel until it was just recessed within the medial intercondylar surface. In both groups, tibial fixation was identical with a bioabsorbable interference screw (BioComposite Screw, Arthrex, North Naples, FL, USA or Milagro screw) and a backup knotless anchor (4.5 mm Biomet Peek knotless anchor, Biomet, Warsaw, IN, USA). The graft was fixed at near full extension after having cycled the knee through range of motion with the graft tensioned.

All patients underwent a specified ACL post-operative rehabilitation protocol depending on concomitant pathology. Cycling was permitted at the six-week mark. In-line jogging typically was allowed at four months with initiation of pivoting motions at seven to eight months. Full return to sports was allowed after nine months. Younger patients enrolled in a sports metrics program followed by a functional ACL exam prior to return to sports. A commuted tomography (CT) scan of the operative knee was obtained postoperatively at six months.

Demographic data including age, gender, and body mass index were collected. The primary outcome measure was bony incorporation of the bone block within the femoral tunnel with CT scan. This was assessed with the femoral ossification score as determined by three board certified radiologists.

The femoral ossification score was devised as a practical means of semi-quantitatively assessing the degree of bone incorporation around the femoral bone plug or screw fixation device present in each patient.

Each CT scan score assessment was performed by one of three musculoskeletal fellowship-trained radiologists. Whenever an ossification score was deemed to be borderline between two categories, a consensus score was determined by two of the radiologists. The impression in the CT report included the femoral ossification score as well as a footnote with the entire scale to explain the score.

Secondary outcome measures included pain score on a visual analogue scale (VAS) obtained preoperatively, at the first post-operative visit, and at return to sports. Physical examination findings included range of motion (ROM) and Lachman grading which were measured preoperatively and at return to sporting activities. Finally, the International Knee Documentation Committee (IKDC) subjective knee evaluation score, Tegner-Lysholm Knee score, and Cincinnati Knee Rating system scores were assessed both pre-operatively and post-operatively at return to sports.

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 18 and 50 able to provide informed consent with ACL tears meeting the indications for reconstruction and electing to undergo reconstruction with an Achilles tendon allograft.

Exclusion Criteria:

* History of prior ACL reconstruction
* pregnancy
* inflammatory disease
* a primary bone disorder
* those taking bone resorption inhibitor medications
* those with injuries to the collateral ligaments or posterior cruciate ligament

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Femoral Ossification Score | 6 months post-op
  Amount of ossification (osseous integration) around the graft at 6 months post-operatively as seen on CT scan. Score range: 0 (minimum) - 5 (maximum). Score of 0 is the worst outcome and indicates no ossification in the femoral tunnel as seen on CT scan. Score of 5 indicates full ossification of the tunnel (best outcome) as seen on CT scan. Scores in between indicate partial ossification (each number 20% more ossification than the previous score).

SECONDARY OUTCOMES:
Pain (VAS) | Obtained preoperatively (right before surgery); 2 weeks after surgery; and 6 months after surgery
  Pain as assessed by the visual analog scale. Scale of 0-10 (0 is the best [no pain], 10 is the worst [severe pain])
Knee range of motion | Obtained preoperatively (right before surgery) and at 6 months after surgery
  Knee range of motion (measured in degrees [angle] from full extension to full flexion). 0 degrees is considered full extension. 140 degrees is full flexion.
International Knee Documentation Committee (IKDC) subjective knee score | Obtained preoperatively (right before surgery) and at 6 months after surgery
  The IKDC is a patient-completed tool, which contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Anup Shah, Principal Investigator — Kelsey-Seybold Clinic
Locations (1):
- Kelsey-Seybold Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Primary and secondary outcome measures (de-identified)
Supporting Information: Study Protocol, CSR
Time Frame: Data is already available (study has been completed)
Access Criteria: Standard